CLINICAL TRIAL: NCT03780192
Title: INSPIRON Sirolimus Eluting Stent Performance in Bifurcation Coronary Arteries Treated Using Provisional Technique
Acronym: insProvisional
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Principal Investigator, Marco Vugman Wainstein, Principal Investigator Hospital Moinhos de Vento, Scitech Produtos Medicos Ltda
Other Study IDs: SC-INS-001-2019
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Bifurcation Lesion; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Bifurcation lesion treatment using provisional stent technique
  Interventions: Device: Inspiron Sirolimus Eluting Stent

INTERVENTIONS:
Device: Inspiron Sirolimus Eluting Stent — Bifurcation treatment using provisional stent technique

SUMMARY:
Evaluate the efficacy of the Inspiron Sirolimus Eluting Stent on bifurcation coronary artery lesions, in order to preserve and not compromize the side branch using the provisional stent technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease on bifurcation anatomy with indication of drug eluting stent implantation , on which the side branch is ≥ 2.5 mm diameter and ostial stenosis ≤50% (Medina 1-1-0, 1-0-0, 0-1-0).

Exclusion Criteria:

* Acute Myocardial Infarction (STMI);
* Chronic occlusion;
* Cardiogenic shock;
* Ejection fraction ≤ 20%;
* Thrombocytopenia (≤ 50 mil);
* DAPT contraindication;
* Life expectancy of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with bifurcation coronary artery disease with indication for drug eluting implantation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Stenosis | day 0
  % of stenosis on side branch after stent placement on main vessel

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No